CLINICAL TRIAL: NCT03992651
Title: Validation of Optical Transcutaneous Sensors to Measure Capnia and Tissue Oxygenation
Brief Title: Optical Transcutaneous Sensors of Capnia and Oxygenation
Acronym: CTCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EssaiClinique_CTCO
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Intervention Model Description: One single group will have simultaneous measurements of capnia and tissue oxygenation by the new sensors and by the standard laboratory sensors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): One single group of healthy subjects
  Interventions: Device: Measurements of capnia and tissue oxygenation by optical transcutaneous sensors

INTERVENTIONS:
Device: Measurements of capnia and tissue oxygenation by optical transcutaneous sensors — Capnia and tissue oxygenation will be measured by optical transcutaneous sensors

SUMMARY:
This study aims at validating new optical transcutaneous sensors to evaluate tissue capnia (CO2 partial pressure) and oxygenation (blood oxygen saturation) by comparing them to standard laboratory measurements (end tidal CO2 measurements and oxygen saturation by near-infrared spectroscopy).

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 50 year old
* Individual having health insurance
* Individual able to provided informed consent
* Subjects with no known pathology and not taking any medical treatment a priori capable of interfering with controlled hypoxia at levels required in the protocol

Exclusion Criteria:

* Body mass index >27 kg/m²
* History of acute mountain sickness
* Chronic diseases know to be associated with high methemoglobinemia
* Known allergy to one of the materials used in the devices (lycra, polyamide...), or to the adhesive plaster.
* Active smoker (>3 cigarets/day)
* Alcohol consumption (>10g/day)
* Individual with high skin sensitivity due to skin diseases
* Mental disorders
* Persons who refuse to sign the information sheet and participation agreement
* Persons under guardianship or not subject to a social security system
* Pregnant woman, parturient, breastfeeding mother
* Person deprived of liberty by judicial or administrative decision
* A person who is subject to a legal protection measure that cannot be included in clinical trials.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Comparison of capnia values | Continuous measurement during the only experimental session (1 hour)
  Comparison of capnia values measured by the new sensors and the standard laboratory sensors

SECONDARY OUTCOMES:
Comparison of tissue oxygenation values | Continuous measurement during the only experimental session (1 hour)
  Comparison of tissue oxygenation values measured by the new sensors and the standard laboratory sensors

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Doutreleau, MD PhD, Principal Investigator — Grenoble Alpes Hospital
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koenig A, Petitdidier N, Grateau H, Characoun S, Ghaith A, Verges S, Doutreleau S, Gharbi S, Gerbelot R, Gioux S, Dinten JM. Contact, high-resolution spatial diffuse reflectance imaging system for skin condition diagnosis: a first-in-human clinical trial. J Biomed Opt. 2021 Jan;26(1):012706. doi: 10.1117/1.JBO.26.1.012706. PMID 33515218